CLINICAL TRIAL: NCT03487653
Title: Detection of the Most Common Micro Organism of Infective Endocarditis in Assiut University Hospital
Brief Title: Detection of the Most Common Microorganism of Infective Endocarditis in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Safaa Samir (Other)
Responsible Party: Sponsor-Investigator, Safaa Samir, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Assiut university hosbital
Record Dates: First submitted 2018-03-01; First posted 2018-04-04 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-03

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: microbiology:Blood culture and sensitvity test .Serology — Gram stain ,Blood culture ,sensitivity test ,biochemical reactions and serological study will be done

SUMMARY:
Indocarditis is an endogenous infection acquired when organisms entering the blood

stream establish on the heart valves, therefore, any bacteremia can potentially result in endocarditis.

Infective endocarditis is an uncommon disease that often presents as pyrexia of unknown origin.

The mortality rate in endocarditis was very high before the antibiotic era, even now a day, the

mortality rate is around 20%(1).A variety of microorganisms can cause IE; staphylococci and streptococci account for the majority of cases. Staphylococcal IE is a common cause of healthcare-associated IE ; streptococcal IE is a common cause of community-acquired IE. Common bacterial pathogens include Staphylococcus aureus , Viridans group streptococci , Enterococcus, Coagulase-negative staphylococci , Streptococcus bovis , other streptococci , gram-negative bacteria, HACEK organisms in this category include a number of fastidious gram-negative bacilli: Haemophilus aphrophilus(subsequently called Aggregatibacter aphrophilus and Aggregatibacter paraphrophilus); Actinobacillus actinomycetemcomitans (subsequently called Aggregatibacter actinomycetemcomitans); Cardiobacterium hominis; Eikenella corrodens; and Kingella kingae , and fungi (1,2). A variable proportion of IE remain blood culture- negative (1-4). Most clinically significant bacteremias are detected within 48 hours; common and fastidious pathogens (such as members of the HACEK group) may be detected within five days of incubation with modern automated blood culture detection systems. The optimal volume of blood for each blood culture in adults is 20 ml.

Zoonotic agents, such as Coxiella burnetii, Brucella spp., and Bartonella spp. were frequently detected in North Africa and identified as causes of infective endocarditis (IE) in Egypt (3,4).Blood culture is the most important investigation for diagnosing infective endocarditis

andto know the prevalence rate of different bacteria and their antibiotic sensitivity pattern.Positive blood culture is the cornerstone of microbiological diagnosis of IE; three sets of blood cultures detect 96 to 98 percent of bacteremia. At least three sets of blood cultures should be obtained from separate venipuncture sites prior to initiation of antibiotic therapy. Patients with IE typically have continuous bacteremia; therefore, blood cultures may be collected at any time and need not necessarily be obtained at the time of fever or chills.

MATERIAL and METHOD A total of 150 blood cultures were received from 50 clinically diagnosed cases of bacterial endocarditis .

Blood sample was collected under all aseptic precautions.

ELIGIBILITY:
Inclusion Criteria:patients that are clinically diagnosed as infective endocarditis before starting antibiotics

Exclusion Criteria:patients that receive antibiotics before taking the blood sample

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Detection of the most common organism of infective endocarditis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Detection of the most common micro organism of infective endocarditis | 2years
  Detection of the most common microorganism of infective endocarditis

IPD SHARING:
Plan to Share IPD: Undecided